CLINICAL TRIAL: NCT00676520
Title: XIENCE V® Everolimus Eluting Coronary Stent System (EECSS) USA Post-Approval Study
Brief Title: XIENCE V® Everolimus Eluting Coronary Stent System USA Post-Approval Study (XIENCE V® USA-Phase 1)
Acronym: XVU-Phase 1
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 06-374
Record Dates: First submitted 2007-10-16; First posted 2008-05-13 (Estimated); Results first posted 2012-11-20 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-10

CONDITIONS: Coronary Artery Disease
Keywords: Angioplasty; Coronary Restenosis; Coronary Artery Disease; Coronary Artery Restenosis; Coronary Artery Stenosis; Total Artery Occlusion; Stents; Stent Thrombosis; Total Coronary Occlusion; Vascular Disease; Myocardial Ischemia
MeSH Terms: conditions — Coronary Artery Disease; Coronary Restenosis; Coronary Stenosis; Vascular Diseases; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Single-arm study
  Interventions: Device: XIENCE V® Everolimus Eluting Coronary Stent

INTERVENTIONS:
Device: XIENCE V® Everolimus Eluting Coronary Stent — Single-arm study designed to evaluate XIENCE V® EECSS continued safety and effectiveness during commercial use in real world settings.

SUMMARY:
XIENCE V USA is a prospective, multi-center, multi-cohort post-approval study. The objectives of this study are

* To evaluate XIENCE V EECSS continued safety and effectiveness during commercial use in real world settings, and
* To support the Food and Drug Administration (FDA) dual antiplatelet therapy (DAPT) initiative. This initiative is designed to evaluate the composite of all death, myocardial infarction (MI) and stroke (MACCE) and the survival of patients that are free from Academic Research Consortium (ARC) definite or probable stent thrombosis (ST) and that have been treated with drug eluting stents (DES) and extended dual antiplatelet therapy.

DETAILED DESCRIPTION:
Study Phase I is from index procedure to 1 year. This prospective, open-label, multi-center, observational, single-arm study is designed to evaluate XIENCE V EECSS safety and effectiveness in real world settings up to 1 year after implantation. The primary endpoint is the stent thrombosis (definite and probable) rate up to 1 year as ARC. The co-primary endpoint is the composite rate of cardiac death and any MI at 1 year. Up to 8,000 patients are planned to be consecutively enrolled at up to 275 sites in the U.S. Clinical follow-up will occur at 14, 30, 180 days and 1 year.

All patients enrolled in the XIENCE V USA who have completed Study Phase I will be evaluated at 1 year to determine whether they are eligible to participate in one of the following cohorts in Study Phase II: XIENCE V USA Long Term Follow-up (LTF) Cohort, Harvard Clinical Research Institute (HCRI) DAPT Cohort, or Abbott Vascular (AV) DAPT Cohort.

ELIGIBILITY:
Inclusion Criteria:

* The patient agrees to participate in this study by signing the Institutional Review Board approved informed consent form.

Exclusion Criteria:

* The inability to obtain an informed consent.

Age limit is determined by investigator.

There are no angiographic inclusion or exclusion criteria for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who agree to participate by signing the Institutional Review Board (IRB) approved informed consent form, and who recieve only XIENCE V® EECSS during the index procedure.
Sampling Method: Non-Probability Sample
Enrollment: 8053 (Actual)
Dates: Start 2008-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Hermiller, MD, Principal Investigator — Heart Center of Indianapolis; Mitch Krucoff, MD, Principal Investigator — Duke University
Locations (1):
- Abbott Vascular, Santa Clara, California, United States

REFERENCES:
- [Derived] Genereux P, Rutledge DR, Palmerini T, Caixeta A, Kedhi E, Hermiller JB, Wang J, Krucoff MW, Jones-McMeans J, Sudhir K, Simonton CA, Serruys PW, Stone GW. Stent Thrombosis and Dual Antiplatelet Therapy Interruption With Everolimus-Eluting Stents: Insights From the Xience V Coronary Stent System Trials. Circ Cardiovasc Interv. 2015 May;8(5):e001362. doi: 10.1161/CIRCINTERVENTIONS.114.001362. PMID 25940520
- [Derived] Sudhir K, Hermiller JB, Naidu SS, Henry TD, Mao VW, Zhao W, Ferguson JM, Wang J, Jonnavithula L, Simonton CA, Rutledge DR, Krucoff MW; XIENCE V USA Investigators. Clinical outcomes in real-world patients with acute myocardial infarction receiving XIENCE V(R) everolimus-eluting stents: one-year results from the XIENCE V USA study. Catheter Cardiovasc Interv. 2013 Oct 1;82(4):E385-94. doi: 10.1002/ccd.24749. Epub 2013 Mar 28. PMID 23172848
- [Derived] Hermiller JB, Rutledge DR, Gruberg L, Katopodis JN, Lombardi W, Mao VW, Zhao W, Sharma SK, Tamboli HP, Wang J, Jonnavithula L, Sudhir K, Krucoff MW. Sustained low clinical event rates in real-world patients receiving everolimus-eluting coronary stent system from a large, prospective, condition of approval study: 2-year clinical outcomes from the XIENCE V USA Study. J Interv Cardiol. 2012 Dec;25(6):565-75. doi: 10.1111/j.1540-8183.2012.00766.x. Epub 2012 Sep 23. PMID 22998355
- [Derived] Naidu SS, Krucoff MW, Rutledge DR, Mao VW, Zhao W, Zheng Q, Wilburn O, Sudhir K, Simonton C, Hermiller JB. Contemporary incidence and predictors of stent thrombosis and other major adverse cardiac events in the year after XIENCE V implantation: results from the 8,061-patient XIENCE V United States study. JACC Cardiovasc Interv. 2012 Jun;5(6):626-35. doi: 10.1016/j.jcin.2012.02.014. PMID 22721657
- [Derived] Krucoff MW, Rutledge DR, Gruberg L, Jonnavithula L, Katopodis JN, Lombardi W, Mao VW, Sharma SK, Simonton CA, Tamboli HP, Wang J, Wilburn O, Zhao W, Sudhir K, Hermiller JB. A new era of prospective real-world safety evaluation primary report of XIENCE V USA (XIENCE V Everolimus Eluting Coronary Stent System condition-of-approval post-market study). JACC Cardiovasc Interv. 2011 Dec;4(12):1298-309. doi: 10.1016/j.jcin.2011.08.010. PMID 22192371

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects are derived from the USA interventional cardiology population.
Pre-assignment Details: A sub-set of subjects was randomized to the DAPT portion of this study.
Period: Overall Study
Arm/Group | Subjects Receiving the XIENCE V EECSS
Started | 8040
Completed | 7309
Not Completed | 731
Not completed — Withdrawal by Subject | 163
Not completed — Lost to Follow-up | 162
Not completed — Death | 159
Not completed — Physician Decision | 20
Not completed — Ineligible for Randomization to DAPT | 209
Not completed — Other Reason | 18

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 8040
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4121
  >=65 years | 3919
Age Continuous [Mean (Standard Deviation); unit: years] | 64.58 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2441
  Male | 5599
Region of Enrollment [Number; unit: participants]
  United States | 8040

OUTCOME MEASURES:

1. Primary Outcome: Stent Thrombosis (Definite and Probable) Rate as Defined by ARC (Academic Research Constortium).
Description: ARC Defines Stent Thrombosis in the following way:
  Definite Stent Thrombosis: Angiographic or pathologic confirmation of partial or total thrombotic occlusion within the peri-stent region AND at least ONE of the following, additional criteria:
  Acute ischemic symptoms Ischemic ECG changes Elevated cardiac biomarkers
  Probable Stent Thrombosis: Any unexplained death within 30 days of stent implantation or any myocardial infarction, which is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause
  Possible Stent Thrombosis Any unexplained death beyond 30 days
  For further information on ARC definitions, please refer to the following website: http://circ.ahajournals.org/content/115/17/2344.full#sec-1
Time Frame: up to 1 year
Population: Enrolled population is defined in the protocol as patients who received only XIENCE V EECSS during the index procedure. First Enrollment Phase and Second Enrollment Phase Pooled.
  The analysis population at clinical follow-up visits may have changed due to early termination from the study by the patient or physician.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7380
percentage of participants | 0.81 [0.62 to 1.05]

2. Primary Outcome: Composite Rate of Cardiac Death and Any Myocardial Infarction (MI)
Description: MI= ARC (Academic Research Constortium) defined
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7522
percentage of participants | 7.2 [6.67 to 7.85]

3. Secondary Outcome: Clinical Device Success
Time Frame: acute: post index procedure until hospital discharge
Population: Enrolled population is defined in the protocol as patients who received only XIENCE V EECSS during the index procedure. First Enrollment Phase and Second Enrollment Phase Pooled.
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 8040
Number analyzed (Lesions) | 11049
percentage of lesions | 99.8 [99.73 to 99.90]

4. Secondary Outcome: Procedural Success
Time Frame: acute: post index procedure until hospital discharge
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 8002
percentage of participants | 97.3 [96.87 to 97.60]

5. Secondary Outcome: Composite Rate of Cardiac Death and Any MI (Q-wave and Non Q-wave)
Description: MI= Academic Research Consortium (ARC) defined
Time Frame: at 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7963
percentage of participants | 3.6 [3.19 to 4.02]

6. Secondary Outcome: Composite Rate of Cardiac Death and Any MI (Q-wave and Non Q-wave)
Description: MI= Academic Research Consortium (ARC) defined
Time Frame: at 180 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7854
percentage of participants | 5.4 [4.88 to 5.89]

7. Secondary Outcome: Composite Rate of All Death and Any MI (Q-wave and Non Q-wave)
Description: MI= Academic Research Consortium (ARC) defined
Time Frame: at 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7963
percentage of participants | 3.6 [3.23 to 4.06]

8. Secondary Outcome: Composite Rate of All Death and Any MI (Q-wave and Non Q-wave)
Description: MI= Academic Research Consortium (ARC) defined
Time Frame: at 180 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7854
percentage of participants | 5.8 [5.34 to 6.39]

9. Secondary Outcome: Composite Rate of All Death and Any MI (Q-wave and Non Q-wave)
Description: MI= Academic Research Consortium (ARC) defined
Time Frame: at 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7522
percentage of participants | 8.3 [7.67 to 8.93]

10. Secondary Outcome: Composite Rate of All Death, Any MI (Q-wave and Non Q-wave) and Any Repeat Revascularization (Percutaneous Coronary Intervention [PCI] and Coronary Artery Bypass Graft [CABG])
Description: MI= Academic Research Consortium (ARC) defined
Time Frame: at 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7963
percentage of participants | 4.3 [3.82 to 4.72]

11. Secondary Outcome: Composite Rate of All Death, Any MI (Q-wave and Non Q-wave) and Any Repeat Revascularization (Percutaneous Coronary Intervention [PCI] and Coronary Artery Bypass Graft [CABG])
Description: MI= Academic Research Consortium (ARC) defined
Time Frame: at 180 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7854
percentage of participants | 9.4 [8.77 to 10.08]

12. Secondary Outcome: Composite Rate of All Death, Any MI (Q-wave and Non Q-wave) and Any Repeat Revascularization (Percutaneous Coronary Intervention [PCI] and Coronary Artery Bypass Graft [CABG])
Description: MI= Academic Research Consortium (ARC) defined
Time Frame: at 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7522
percentage of participants | 14.9 [14.11 to 15.73]

13. Secondary Outcome: Composite Rate of Cardiac Death, Any MI (Q-wave and Non Q-wave) Attributed to the Target Vessel, and Target Lesion Revascularization (TLR) (PCI and CABG)
Description: MI= Academic Research Consortium (ARC) defined
Time Frame: at 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7963
percentage of participants | 3.5 [3.10 to 3.92]

14. Secondary Outcome: Composite Rate of Cardiac Death, Any MI (Q-wave and Non Q-wave) Attributed to the Target Vessel, and Target Lesion Revascularization (TLR) (PCI and CABG)
Description: MI= Academic Research Consortium (ARC) defined
Time Frame: at 180 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7854
percentage of participants | 6.3 [5.81 to 6.90]

15. Secondary Outcome: Composite Rate of Cardiac Death, Any MI (Q-wave and Non Q-wave) Attributed to the Target Vessel, and Target Lesion Revascularization (TLR) (PCI and CABG)
Description: MI= Academic Research Consortium (ARC) defined
Time Frame: at 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7522
percentage of participants | 9.6 [8.97 to 10.31]

16. Secondary Outcome: Death (Cardiac Death, Vascular Death, and Non-cardiovascular Death)
Time Frame: at 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7963
percentage of participants | 0.4 [0.23 to 0.51]

17. Secondary Outcome: Death (Cardiac Death, Vascular Death, and Non-cardiovascular Death)
Time Frame: at 180 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7854
percentage of participants | 1.4 [1.13 to 1.66]

18. Secondary Outcome: Death (Cardiac Death, Vascular Death, and Non-cardiovascular Death)
Time Frame: at 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7522
percentage of participants | 2.6 [2.23 to 2.96]

19. Secondary Outcome: Any MI (Q-wave and Non Q-wave)
Description: MI= Academic Research Consortium (ARC) defined
Time Frame: at 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7963
percentage of participants | 3.3 [2.96 to 3.76]

20. Secondary Outcome: Any MI (Q-wave and Non Q-wave)
Description: MI= Academic Research Consortium (ARC) defined
Time Frame: at 180 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7854
percentage of participants | 4.7 [4.28 to 5.23]

21. Secondary Outcome: Any MI (Q-wave and Non Q-wave)
Description: MI= Academic Research Consortium (ARC) defined
Time Frame: at 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7522
percentage of participants | 6.3 [5.78 to 6.89]

22. Secondary Outcome: Revascularization (Target Lesion, Target Vessel [TVR], and Non-target Vessel) (PCI and CABG)
Time Frame: at 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7963
percentage of participants | 1.1 [0.86 to 1.33]

23. Secondary Outcome: Revascularization (Target Lesion, Target Vessel [TVR], and Non-target Vessel) (PCI and CABG)
Time Frame: at 180 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7854
percentage of participants | 5.0 [4.53 to 5.51]

24. Secondary Outcome: Revascularization (Target Lesion, Target Vessel [TVR], and Non-target Vessel) (PCI and CABG)
Time Frame: at 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7522
percentage of participants | 9.2 [8.54 to 9.86]

25. Secondary Outcome: Major Bleeding Complications
Description: by TIMI flow
Time Frame: at 14 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7990
percentage of participants | 0.6 [0.45 to 0.81]

26. Secondary Outcome: Major Bleeding Complications
Description: by TIMI flow
Time Frame: at 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7944
percentage of participants | 0.7 [0.53 to 0.91]

27. Secondary Outcome: Major Bleeding Complications
Description: by TIMI flow
Time Frame: at 180 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7763
percentage of participants | 1.8 [1.47 to 2.07]

28. Secondary Outcome: Major Bleeding Complications
Description: by TIMI flow
Time Frame: at 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7346
percentage of participants | 2.8 [2.40 to 3.16]

29. Secondary Outcome: Dual Antiplatelet Medication Usage
Description: Patient is included if medications (both aspirin and thienopyridine) were taken for at least 1 day during the visit window. The visit window for 14-day visit is 7-21 days, 30-day visit is 23-37 days, 180-day visit is 166-194 days, 1-year visit is 323-407 days, and 2-year visit is 688-772 days.
  Adjunctive antiplatelet therapy includes: Aspirin & Thienopyridines (Clopidogrel/Ticlopidine/Prasugrel).
  Compliance refers to subjects following prescribed instructions for taking these medications. Therapy interruptions refer to any intervals during which the subject stops taking one or all of the prescribed medications.
Time Frame: at 14 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 8039
percentage of participants | 89.4 [88.67 to 90.03]

30. Secondary Outcome: Dual Antiplatelet Medication Usage
Description: as for outcome 29
Time Frame: at 30 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 8039
percentage of participants | 89.2 [88.45 to 89.82]

31. Secondary Outcome: Dual Antiplatelet Medication Usage
Description: as for outcome 29
Time Frame: at 180 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 8039
percentage of participants | 86.4 [85.60 to 87.11]

32. Secondary Outcome: Dual Antiplatelet Medication Usage
Description: as for outcome 29
Time Frame: at 1 year
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 8039
percentage of participants | 79.9 [79.03 to 80.79]

33. Secondary Outcome: Dual Antiplatelet Therapy Non-compliance Through 1 Year
Description: Defined as patients who had at least 1 day without using either aspirin or thienopyridine from 1 to 407 days post index procedure.
Time Frame: 1 year
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 6886
percentage of participants | 18.0

34. Secondary Outcome: Composite Rate of Cardiac Death and MI (Q-wave and Non Q-wave) Attributed to the Target Vessel, and Clinically-indicated Target Lesion Revascularization (CI-TLR) (PCI and CABG) (This Composite Endpoint is Also Denoted as TLF)
Description: MI= Academic Research Consortium (ARC) defined
Time Frame: at 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7963
percentage of participants | 3.5 [3.06 to 3.88]

35. Secondary Outcome: Composite Rate of Cardiac Death and MI (Q-wave and Non Q-wave) Attributed to the Target Vessel, and Clinically-indicated Target Lesion Revascularization (CI-TLR) (PCI and CABG) (This Composite Endpoint is Also Denoted as TLF)
Description: MI= Academic Research Consortium (ARC) defined
Time Frame: at 180 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7854
percentage of participants | 6.2 [5.71 to 6.80]

36. Secondary Outcome: Composite Rate of Cardiac Death and MI (Q-wave and Non Q-wave) Attributed to the Target Vessel, and Clinically-indicated Target Lesion Revascularization (CI-TLR) (PCI and CABG) (This Composite Endpoint is Also Denoted as TLF)
Description: MI= Academic Research Consortium (ARC) defined
Time Frame: at 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 7522
percentage of participants | 9.4 [8.75 to 10.08]

37. Secondary Outcome: Patient Health Status, Physical Limitations Assessed Using the SAQ (Seattle Angina Questionaire)
Description: SAQ: 19-item, 5-6-point Likert, questionnaire measuring 5 dimensions of coronary artery disease:
  Anginal Stability: whether a patient's symptoms are changing over time. Anginal Frequency: how often a patient is having symptoms now Physical Limitation: how much a patient's condition is hampering his ability to do what he wants to do.
  Treatment Satisfaction: how well a patient understands her care and what she thinks of it.
  Disease Perception: the overall impact of a patient's condition on a patient's interpersonal relationships and state of mind.
  Each dimension is assigns each response an ordinal value, beginning with 1 for the response at the lowest level of functioning, and summing across items within each of the 5 scales. Scale scores then transformed to 0-100 range by subtracting the lowest possible scale score, dividing by the range of the scale and multiplying by 100.
Time Frame: at baseline
Population: First enrollment phase of ~5,000 patients only. Enrolled population is defined in the protocol as patients who received only XIENCE V EECSS during the index procedure.
  The analysis population at clinical follow-up visits may have changed due to early termination from the study by the patient or physician.
Measure: Mean (Standard Deviation); unit: units on the SAQ scale
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 4483
units on the SAQ scale | 70.0 (25.5)

38. Secondary Outcome: Patient Health Status, Physical Limitations Assessed Using the SAQ (Seattle Angina Questionaire)
Description: as for outcome 37
Time Frame: at 180 days
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: units on the SAQ scale
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 3648
units on the SAQ scale | 75.8 (24.9)

39. Secondary Outcome: Patient Health Status, Physical Limitations Assessed Using the SAQ (Seattle Angina Questionaire)
Description: as for outcome 37
Time Frame: at 1 year
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: units on the SAQ scale
Arm/Group | Subjects Receiving the XIENCE V EECSS
Number analyzed (Participants) | 3457
units on the SAQ scale | 76.0 (24.9)

40. Secondary Outcome: SAQ (Seattle Angina Questionaire)
Description: as for outcome 37
Time Frame: at baseline
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: units on the SAQ scale
Arm/Group | Physical Limitations | Angina Stability | Angina Frequency | Treatment Satisfaction | Perception of Disease/Quality of Life
Number analyzed (Participants) | 4483 | 4681 | 4767 | 4736 | 4661
units on the SAQ scale | 70.0 (25.5) | 42.0 (27.6) | 73.1 (25.1) | 98.1 (12.7) | 55.3 (25.8)

41. Secondary Outcome: SAQ (Seattle Angina Questionaire)
Description: as for outcome 37
Time Frame: 180 days
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: units on the SAQ scale
Arm/Group | Physical Limitations | Angina Stability | Angina Frequency | Treatment Satisfaction | Perception of Disease/Quality of Life
Number analyzed (Participants) | 3648 | 3896 | 3903 | 3839 | 3773
units on the SAQ scale | 75.8 (24.9) | 57.3 (20.2) | 90.1 (17.1) | 91.4 (14.5) | 76.8 (21.5)

42. Secondary Outcome: SAQ (Seattle Angina Questionaire)
Description: as for outcome 37
Time Frame: 1 year
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: units on the SAQ scale
Arm/Group | Physical Limitations | Angina Stability | Angina Frequency | Treatment Satisfaction | Perception of Disease/Quality of Life
Number analyzed (Participants) | 3457 | 3689 | 3694 | 3630 | 3574
units on the SAQ scale | 76.0 (24.9) | 54.3 (18.3) | 90.7 (17.0) | 92.2 (14.0) | 78.0 (21.1)

ADVERSE EVENTS:
Time Frame: 1 year
Description: If a subject had more than one event, this subject has been counted only once. The number of participants at risk excludes subjects who were "early terminated" up to 365 days and who had no events through the given timepoint.
Arm/Group | Subjects Receiving the XIENCE V EECSS
Serious Adverse Events (participants affected / at risk) | 1656/4952
Other Adverse Events (participants affected / at risk) | 478/4952
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Receiving the XIENCE V EECSS (N=4952)
Acute coronary syndrome (Cardiac disorders) | 13 (13)
Acute myocardial infarction (Cardiac disorders) | 64 (67)
Acute pulmonary edema (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 510 (632)
Angina unstable (Cardiac disorders) | 50 (57)
Aortic valve disease (Cardiac disorders) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 7 (7)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1)
Arteriospasm coronary (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 51 (58)
Atrial flutter (Cardiac disorders) | 14 (18)
Atrial thrombosis (Cardiac disorders) | 1 (1)
Atrioventricular block (Cardiac disorders) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 16 (16)
Cardiac arrest (Cardiac disorders) | 17 (17)
Cardiac failure (Cardiac disorders) | 14 (16)
Cardiac failure acute (Cardiac disorders) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 83 (120)
Cardiac tamponade (Cardiac disorders) | 4 (4)
Cardio-respiratory arrest (Cardiac disorders) | 9 (9)
Cardiogenic shock (Cardiac disorders) | 6 (6)
Cardiomyopathy (Cardiac disorders) | 9 (9)
Congestive cardiomyopathy (Cardiac disorders) | 2 (2)
Coronary artery dissection (Cardiac disorders) | 14 (14)
Coronary artery disease (Cardiac disorders) | 19 (19)
Coronary artery perforation (Cardiac disorders) | 1 (2)
Coronary artery stenosis (Cardiac disorders) | 4 (4)
Coronary artery thrombosis (Cardiac disorders) | 4 (4)
Electromechanical dissociation (Cardiac disorders) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 4 (4)
Left ventricular dysfunction (Cardiac disorders) | 4 (4)
Low cardiac output syndrome (Cardiac disorders) | 1 (1)
Mitral valve calcification (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 6 (7)
Mitral valve stenosis (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 31 (31)
Myocardial ischaemia (Cardiac disorders) | 14 (15)
Palpitations (Cardiac disorders) | 4 (4)
Pericardial effusion (Cardiac disorders) | 3 (4)
Pericardial haemorrhage (Cardiac disorders) | 1 (1)
Post procedural myocardial infarction (Cardiac disorders) | 3 (3)
Sick sinus syndrome (Cardiac disorders) | 12 (12)
Sinus arrest (Cardiac disorders) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sudden cardiac death (Cardiac disorders) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 4 (4)
Tachycardia (Cardiac disorders) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Ventricular dysfunction (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 9 (9)
Ventricular tachycardia (Cardiac disorders) | 24 (27)
Adverse drug reaction (General disorders) | 2 (2)
Asthenia (General disorders) | 6 (6)
Catheter site haematoma (General disorders) | 16 (16)
Catheter site haemorrhage (General disorders) | 7 (7)
Drug withdrawal syndrome (General disorders) | 1 (1)
Exercise tolerance decreased (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Gait disturbance (General disorders) | 1 (1)
Generalised edema (General disorders) | 1 (1)
Infusion site phlebitis (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 167 (191)
Edema (General disorders) | 2 (2)
Edema peripheral (General disorders) | 5 (5)
Pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 9 (10)
Sudden death (General disorders) | 2 (2)
Systemic inflammatory response syndrome (General disorders) | 1 (1)
Contrast media reaction (Immune system disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2)
Coronary artery reocclusion (Injury, poisoning and procedural complications) | 1 (1)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 2 (2)
Device dislocation (Injury, poisoning and procedural complications) | 1 (1)
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 1 (1)
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 3 (3)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 17 (18)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Lead dislodgement (Injury, poisoning and procedural complications) | 1 (1)
Mechanical complication of implant (Injury, poisoning and procedural complications) | 2 (2)
Other injuries (Injury, poisoning and procedural complications) | 53 (59) — Other injuries consists of all the PTs which were not in Administration site reactions and Procedural and device related injuries HLGT category for the corresponding SOC.
Pacemaker complication (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhagen (Injury, poisoning and procedural complications) | 4 (4)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Reperfusion injury (Injury, poisoning and procedural complications) | 7 (7)
Stent-graft endoleak (Injury, poisoning and procedural complications) | 1 (1)
Thrombosis in device (Injury, poisoning and procedural complications) | 5 (5)
Vessel perforation (Injury, poisoning and procedural complications) | 1 (1)
Weaning failure (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Amnesia (Nervous system disorders) | 2 (2)
Anoxic encephalopathy (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Carotid sinus syndrome (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 23 (24)
Complex partial seizures (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 4 (4)
Dementia (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 20 (20)
Dizziness postural (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 2 (2)
Embolic cerebral infarction (Nervous system disorders) | 1 (1)
Embolic stroke (Nervous system disorders) | 4 (4)
Encephalopathy (Nervous system disorders) | 1 (1)
Facial palsy (Nervous system disorders) | 1 (1)
Facial paresis (Nervous system disorders) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 2 (2)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (5)
Hemiparesis (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 2 (2)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 5 (5)
Hypoglycaemic encephalopathy (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 5 (5)
Lethargy (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Moyamoya disease (Nervous system disorders) | 1 (1)
Muscular weakness (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Neurological symptom (Nervous system disorders) | 1 (1)
Neuromyelitis optica (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 3 (3)
Parkinson's disease (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 7 (7)
Spondylitic myelopathy (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 37 (38)
Syncope vasovagal (Nervous system disorders) | 3 (3)
Tension headache (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 19 (20)
Unresponsive to stimulie (Nervous system disorders) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1)
Vertigo (Nervous system disorders) | 3 (3)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 51 (61)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 2 (2)
Endocrine disorders (Endocrine disorders) | 1 (1)
Eye disorders (Eye disorders) | 5 (5)
Gastrointestinal disorders (Gastrointestinal disorders) | 114 (137)
Hepatobiliary disorders (Hepatobiliary disorders) | 28 (30)
Infections and infestations (Infections and infestations) | 170 (212)
Investigations (Investigations) | 57 (63)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 47 (59)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 58 (63)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 51 (54)
Psychiatric disorders (Psychiatric disorders) | 20 (21)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 3 (4)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 11 (11)
Surgical and medical procedures (Surgical and medical procedures) | 46 (47)
Other renal and urinary disorders (Renal and urinary disorders) | 42 (45) — Other renal and urinary disorders consist of all the PTs which were not in Acute renal failure for the corresponding SOC.
Renal failure acute (Renal and urinary disorders) | 31 (31)
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 31 (34)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 91 (104)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 15 (15)
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Accelerated hypertension (Vascular disorders) | 2 (2)
Aortic aneurysms (Vascular disorders) | 10 (10)
Aortic aneurysm rupture (Vascular disorders) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 4 (4)
Arterial thrombosis limb (Vascular disorders) | 3 (4)
Arteriosclerosis (Vascular disorders) | 9 (9)
Arteriovenous malformation (Vascular disorders) | 1 (1)
Carotid artery disease (Vascular disorders) | 5 (5)
Carotid artery occlusion (Vascular disorders) | 1 (1)
Carotid artery stenosis (Vascular disorders) | 17 (19)
Deep vein thrombosis (Vascular disorders) | 8 (9)
Epistaxis (Vascular disorders) | 3 (3)
Femoral arterial stenosis (Vascular disorders) | 6 (7)
Femoral artery occlusion (Vascular disorders) | 2 (2)
Gastrointestinal haemorrhage (Vascular disorders) | 54 (57)
Haematoma (Vascular disorders) | 3 (3)
Haemoptysis (Vascular disorders) | 4 (4)
Haemorrhage (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 15 (16)
Hypertensive crisis (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 27 (30)
Hypovolaemic shock (Vascular disorders) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 15 (17)
Labile blood pressure (Vascular disorders) | 1 (1)
Muscle haemorrhage (Vascular disorders) | 1 (1)
Oesophageal varices haemorrhage (Vascular disorders) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 4 (4)
Peripheral arterial occlusive disease (Vascular disorders) | 4 (4)
Peripheral ischaemia (Vascular disorders) | 4 (6)
Peripheral vascular disorder (Vascular disorders) | 7 (8)
Pulmonary hypertension (Vascular disorders) | 1 (1)
Rectal haemorrhage (Vascular disorders) | 6 (7)
Renal artery occlusion (Vascular disorders) | 1 (1)
Renal artery stenosis (Vascular disorders) | 9 (9)
Retroperitoneal haemorrhage (Vascular disorders) | 14 (14)
Subclavian artery stenosis (Vascular disorders) | 2 (2)
Thrombosis (Vascular disorders) | 2 (2)
Upper gastrointestinal haemorrhage (Vascular disorders) | 10 (10)
Vascular insufficiency (Vascular disorders) | 1 (1)
Vascular pseudoaneurysm (Vascular disorders) | 18 (18)
Aortic intramural haematoma (Vascular disorders) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Receiving the XIENCE V EECSS (N=4952)
Angina pectoris (Cardiac disorders) | 478 (556)
Non-cardiac chest pain (General disorders) | 280 (325)
Gastrointestinal disorders (Gastrointestinal disorders) | 316 (362)
Infections and infestations (Infections and infestations) | 259 (311)
Investigations (Investigations) | 349 (383)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 459 (535)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days